CLINICAL TRIAL: NCT05164900
Title: Manifestations of Ocular Irritation Following Pterygium Excision With Sutures Fixed Conjunctival Autograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Molham Abdelhafez Elbakary, Assistant professor of Ophthalmology, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 34970/10/21
Record Dates: First submitted 2021-12-04; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Pterygium
Keywords: pterygium excision; conjunctival auto-graft; ocular irritation; conjunctival hyperemia
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with nasal pterygium. (Experimental)
  Interventions: Procedure: pterygium excision with sutures fixed conjunctival auto-graft

INTERVENTIONS:
Procedure: pterygium excision with sutures fixed conjunctival auto-graft — Pterygium excision with vicryl 8/0 fixed conjunctival auto-graft under local anesthesia. During the follow up period, indicators of ocular irritation were assessed.

SUMMARY:
In this work, the manifestations of ocular irritation associated with vicryl 8/0 sutures fixed conjunctival auto-graft in pterygium patients were evaluated. The severity of post-operative foreign body sensation, pain, and watering was subjectively evaluated. The localized nasal quadrant conjunctival hyperemia was also evaluated. It was found that sutures fixed conjunctival auto-graft can be used safely with short-term minimal to moderate tolerable manifestations of ocular irritation with no significant complications.

DETAILED DESCRIPTION:
All the patients were subjected to pterygium excision surgery with conjunctival auto-graft under local anesthesia. The graft was fixed by vicryl 8-0 sutures.Ocular irritation symptoms including pain, foreign body sensation and watering were subjectively evaluated. Pain was evaluated using 5 points scale, where (0) indicated no pain; (1) very mild easily tolerable pain; (2) mild pain with discomfort; (3) moderate pain that interfered with the usual activities; (4) severe pain that totally interfered with performing daily activities or sleep. Foreign body sensation and watering of the eye were evaluated with the use of a 4 points abnormal sensation scale, where (0) indicated no abnormal sensation; (1) is somewhat bothersome; (2) is moderately bothersome; (3) is very bothersome. The score of patients' subjective symptoms evaluation were collected in a total score which ranged from zero to a maximum of 10. A total score of 3 or less was considered as minimal irritation (grade I), 4-6 was considered as mild-moderate tolerable irritation (grade II), and 7 or more was considered as severe annoying irritation (grade III).

The degree of localized conjunctival hyperemia involving the nasal quadrant was evaluated 2 weeks, 1,2 and 3 months post-operative using the Cornea and Contact Lens Research Unit (CCLRU) photographic grading scale. In this scale 1 refers to very slight; 2 slight; 3 moderate; 4 severe. Decimal fraction of 0.5 was added to describe the intermediate cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pterygium

Exclusion Criteria:

* Previous ocular surgeries
* Ocular surface disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Ocular pain was subjectively evaluated. | 1 week after surgery.
  The pain was evaluated using 5 points scale, where (0) indicated no pain; (1) very mild easily tolerable pain; (2) mild pain with discomfort; (3) moderate pain that interfered with the usual activities; (4) severe pain that totally interfered with performing daily activities or sleep.
Change of ocular pain subjective evaluation. | 2 weeks, 1 month, 2 and 3 months post-operative.
  The pain was evaluated using 5 points scale, where (0) indicated no pain; (1) very mild easily tolerable pain; (2) mild pain with discomfort; (3) moderate pain that interfered with the usual activities; (4) severe pain that totally interfered with performing daily activities or sleep.
Ocular foreign body sensation was subjectively evaluated. | 1 week after surgery.
  Foreign body sensation was evaluated with the use of a 4 points abnormal sensation scale, where (0) indicated no abnormal sensation; (1) is somewhat bothersome; (2) is moderately bothersome; (3) is very bothersome.
Change of ocular foreign body sensation subjective evaluation. | 2 weeks, 1 month, 2 and 3 months post-operative.
  Foreign body sensation was evaluated with the use of a 4 points abnormal sensation scale, where (0) indicated no abnormal sensation; (1) is somewhat bothersome; (2) is moderately bothersome; (3) is very bothersome.
Watering of the eye was subjectively evaluated. | 1 week after surgery.
  Watering of the eye was evaluated with the use of a 4 points abnormal sensation scale, where (0) indicated no abnormal sensation; (1) is somewhat bothersome; (2) is moderately bothersome; (3) is very bothersome.
Change of watering of the eye subjective evaluation. | 2 weeks, 1 month, 2 and 3 months post-operative.
  Watering of the eye was evaluated with the use of a 4 points abnormal sensation scale, where (0) indicated no abnormal sensation; (1) is somewhat bothersome; (2) is moderately bothersome; (3) is very bothersome.
The degree of localized conjunctival hyperemia involving the nasal quadrant was evaluated. | 2 weeks after surgery.
  The degree of localized conjunctival hyperemia involving the nasal quadrant was evaluated using the cornea and contact lens research unit (CCLRU) photographic grading scale. In this scale 1 refers to very slight; 2 slight; 3 moderate; 4 severe.
Change of the degree of localized conjunctival hyperemia involving the nasal quadrant was evaluated. | 1month,2 and 3 months post-operative.
  The degree of localized conjunctival hyperemia involving the nasal quadrant was evaluated using the cornea and contact lens research unit (CCLRU) photographic grading scale. In this scale 1 refers to very slight; 2 slight; 3 moderate; 4 severe.

CONTACTS AND LOCATIONS:
Overall Officials: Molham Elbakary, Principal Investigator — Assitant professor of Ophthalmology
Locations (1):
- Faculty of Medicine, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No